CLINICAL TRIAL: NCT04955938
Title: A Phase Ib Study of Fedratinib With IDH Inhibition in Advanced-Phase, IDH-Mutated Ph-Negative Myeloproliferative Neoplasms
Brief Title: A Study of Fedratinib With IDH Inhibition in Advanced-Phase, IDH-Mutated Ph-Negative Myeloproliferative Neoplasms
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: unable to accrue
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB21-0483
Record Dates: First submitted 2021-06-22; First posted 2021-07-09 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: IDH Mutation; IDH1 Mutation; IDH2 Gene Mutation; Blood Cancer; Myeloproliferative Neoplasm
Keywords: Leukemia; myeloid; blood cancer; Myeloproliferative Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms; Myeloproliferative Disorders; Leukemia | interventions — ivosidenib; enasidenib; fedratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A - Participants with IDH1 Mutations (Experimental): After genetic testing, if participants are found to have IDH1 Mutations (a genetic mutation) then they will be assigned to this group and will receive the following study drugs:
  Single agent Phase (Cycles 1-3):
  The initial phase of treatment will consist of 3 cycles (lasting 28 days) of ivosidenib 500mg daily x 28 days
  Combination Phase (Cycle 4 onwards):
  If a participant shows clinical benefit (including their disease stabilizing) following the first 3- cycle phase, he or she may go onto the combination phase. Combination treatment will consist of ivosidenib daily x 28 days along with fedratinib daily x 28 days.
  Interventions: Drug: Ivosidenib; Drug: Fedratinib
- Arm B - Participants with IDH2 Mutations (Experimental): After genetic testing, if participants are found to have IDH2 Mutations (a genetic mutation) then they will be assigned to this group and will receive the following study drugs:
  Single agent Phase (Cycles 1-3):
  The initial phase of treatment will consist of 3 cycles (lasting 28 days) of enasidenib 100mg daily x 28 days
  Combination Phase (Cycle 4 onwards):
  If a participant shows clinical benefit (including their disease stabilizing) following the first 3- cycle phase, he or she may go onto the combination phase.Combination treatment will consist of enasidenib 100mg daily x 28 days along with fedratinib daily x 28 days.
  Interventions: Drug: Enasidenib; Drug: Fedratinib

INTERVENTIONS:
Drug: Ivosidenib — A drug used to treat acute myeloid leukemia that has a mutated (changed) form of a gene called isocitrate dehydrogenase-1 (IDH1).
  Other Names: Tibsovo
  Arms: Arm A - Participants with IDH1 Mutations
Drug: Enasidenib — A drug used to treat acute myeloid leukemia (AML) that has recurred (come back) or has not gotten better after treatment with other anticancer therapy.
  Other Names: IDHIFA
  Arms: Arm B - Participants with IDH2 Mutations
Drug: Fedratinib — This medication is used to treat a certain type of cancer (myelofibrosis). Fedratinib belongs to a class of drugs known as JAK (janus kinase) inhibitors. It works by slowing or stopping the growth of cancer cells.
  Other Names: INREBIC

SUMMARY:
The purpose of this research is to gather information on the safety and effectiveness of fedratinib (a drug called a "jak inhibitor" ) in combination with ivosidenib or enasidenib (two anti-cancer drugs). While all three drugs are FDA-approved for various conditions, the US Food and Drug Administration (FDA) has not approved the combination of these drugs for the treatment of rare blood cancers that present Isocitrate dehydrogenase (IDH) mutations, and therefore these drugs can only be given in a research study.

DETAILED DESCRIPTION:
Doctors leading this study hope to learn about the safety of combining fedratinib (a type of drug called a "JAK inhibitor" whichblocks the activity of janus kinase enzymes in your body) with anti-cancer drugs ivosidenib and enasidenib in participants who have rare blood cancers that show Isocitrate dehydrogenase (IDH) mutations (a type of genetic mutation). Your participation in this research will last about 24 months.

The purpose of this research is to gather information on the safety and effectiveness of fedratinib in combination with ivosidenib or enasidenib. While all three drugs are FDA-approved for various conditions, the US Food and Drug Administration (FDA) has not approved the combination of these drugs for the treatment of IDH-mutated blood cancers (known as myeloproliferative neoplasms), and therefore these drugs can only be given in a research study.

ELIGIBILITY:
Inclusion Criteria:

Must be diagnosed with advanced-Phase IDH-mutated Ph-neg MPNs (both untreated and relapsed/refractory) including any of the following:

* polycythemia vera with (PV) ≥ 5% blasts
* essential thrombocythemia (ET) with ≥ 5% blasts
* primary myelofibrosis (PMF) with ≥ 5% blasts
* Atypical CML with ≥ 5% blasts
* MPN-NOS with ≥ 5% blasts
* MDS/MPN Overlap Syndromes with ≥ 5% blasts including CMML
* post-PV myelofibrosis with ≥ 5% blasts
* post-ET myelofibrosis with ≥ 5% blasts
* Patients can be on cytoreduction at time of study enrollment with hydroxyurea or steroids.
* Age ≥18 years. Because no dosing or adverse event data are currently available on the use of fedratinib in combination with IDH inhibitors in patients <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* Eastern Cooperative Oncology Group performance status ≤2 (see Appendix A).

Patients must have normal organ and marrow function as defined below:

* Creatinine clearance ≥30 mL/min, determined by the Cockroft-Gault formula, OR serum creatinine ≤ 1.5 x ULN
* AST and ALT ≤3 x ULN and bilirubin ≤1.5 x ULN (unless considered due to Gilbert's syndrome, leukemic involvement, or extravascular hemolysis in the spleen)

Other eligibility criteria includes the following:

* Patients must be at least 2 weeks from major surgery, radiation therapy, or participation in other investigational trials, and must have recovered from clinically significant toxicities related to these prior treatments.
* Female patients of childbearing potential must have negative results for a pregnancy test
* Patients must be willing to use appropriate contraception. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria

* Patients cannot be on concomitant chemotherapy, radiation therapy, or immunotherapy other than as specified in this protocol. Patients cannot have had prior treatment with an IDH1 inhibitor, IDH2 inhibitor, or fedratinib.
* Patients with a "currently active" second malignancy other than non-melanoma skin cancers. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are free of disease for ≥ 3 years or they are not currently requiring treatment for an indolent malignancy.
* Patients with prior history of encephalopathy, including Wernicke's (WE). If a patient has signs/symptoms of encephalopathy, including WE (eg severe ataxia, ocular paralysis or cerebellar signs) in which case thiamine deficiency needs to be excluded and a brain MRI might be required to exclude possible Wernicke's encephalopathy. Patients with thiamine deficiency that has not been corrected before proceeding to the dose finding phase of the study
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to fedratinib, ivosidenib, or enasidenib.
* Patients receiving any medications or substances that are inhibitors or inducers of CYP3A4 should have eligibility and alternative medications reviewed by site PI. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list such as http://medicine.iupui.edu/clinpharm/ddis/table.aspx; medical reference texts such as the Physicians' Desk Reference may also provide this information. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, active chronic liver disease (eg chronic alcoholic liver disease, autoimmune hepatitis, sclerosing cholangitis, primary biliary cholangitis, hemochromatosis) or psychiatric illness/social situations that would limit compliance with study requirements.
* Subject has a history of progressive multifocal leukoencephalopathy (PML)
* Subject has QTc interval (ie, Fridericia's correction [QTcF]) ≥ 450 msec or other factors that increase the risk of QT prolongation or arrhythmic events (e.g. family history of long QT interval syndrome) at screening unless due to bundle branch block or pacemaker with approval of the principal investigator.
* Pregnant women are excluded from this study because fedratinib, ivosidenib, and enasidenib carry the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with fedratinib, ivosidenib, and enasidenib, breastfeeding should be discontinued if the mother is treated with any of these agents.
* HIV-positive patients, patients with active hepatitis B, and patients with active Hepatitis C on antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with fedratinib, ivosidenib, and enasidenib. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Patient is known to have dysphagia, short-gut syndrome, gastroparesis, or other conditions that limit the ingestion or gastrointestinal absorption of drugs administered orally.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-06-07 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of Fedratinib Combined with Ivosidenib in Participants Who Have IDH1 Mutations | 24 months
  The maximum tolerated dose of fedratinib in combination with ivosidenib in participants who have IDH1-mutated blood cancer. This will be assessed by the number of reported dose-limiting toxicities and adverse events among participants according to the Common Terminology Criteria for Adverse Events version 5.
Maximum Tolerated Dose of Fedratinib Combined with Enasidenib in Participants Who Have IDH2 Mutations | 24 months
  The maximum tolerated dose of fedratinib in combination with ivosidenib in participants who have IDH1-mutated blood cancer. This will be assessed by the number of reported dose-limiting toxicities and adverse events among participants according to the Common Terminology Criteria for Adverse Events version 5.

SECONDARY OUTCOMES:
1-Year Overall Survival | 12 months
  The number of patients who are living 1 year after the beginning of treatment on study as assessed by data from clinical records.
Overall Response Rate (ORR) | 24 months
  Overall response rate as assessed by the number of participants who achieve a complete molecular response (CMR), cytogenetic complete response (CCR), acute leukemia response-complete (ALR-C), or acute leukemia response-partial (ALR-P).
Time to Response | 24 months
  Time to response will be defined as time from treatment administration to first documented complete molecular response (CMR), cytogenetic complete response (CCR), acute leukemia response-complete (ALR-C), or acute leukemia response-partial (ALR-P). DCR will be defined as the portion of subjects achieving a complete molecular response,cytogenetic complete response (CCR), acute leukemia response-complete (ALR-C), or acute leukemia response-partial (ALR-P) or stabilized disease for ≥ 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Olatoyosi Odenike, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided